CLINICAL TRIAL: NCT04288258
Title: A Health and Wellness Lifestyle Program to Support Community-Dwelling Persons With Traumatic Brain Injury (TBI) and Their Caregivers: In-House Research Project, Objective 2
Brief Title: A Health and Wellness Lifestyle Program to Support Community-Dwelling Persons With Traumatic Brain Injury
Acronym: POWERS-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura E. Dreer, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90DPTB0015
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: case-control crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Health and Wellness Program
  Interventions: Behavioral: Telehealth-Based Health and Wellness Program (POWERS-TBI)

INTERVENTIONS:
Behavioral: Telehealth-Based Health and Wellness Program (POWERS-TBI) — The treatment program is interactive and will be delivered via the internet, along with ongoing telephone health coaching calls designed to motivate, problem-solve challenges, reinforce skills learned, and prevent relapse.

SUMMARY:
To evaluate the efficacy of an adapted telehealth-based, health and wellness lifestyle program on promoting healthy lifestyle behaviors and improving health outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of an adapted telehealth-based, health and wellness lifestyle program (POWERS-TBI) on promoting healthy lifestyle behaviors and improving self-efficacy for healthy activities such as amount of physical activity, dietary/food intake, mental stimulation and activity, substance use, mindfulness/spirituality, social relationships, and/or leisure activities among persons with TBI and their caregivers. The treatment program will be delivered via the internet, along with ongoing telephone health coaching calls designed to motivate, problem-solve challenges, reinforce skills learned, and prevent relapse. The goals are to evaluate the impact of the treatment program on improving health outcomes for people with TBI. The investigators plan to accomplish this by evaluating the impact of the program using a case-control crossover design.

ELIGIBILITY:
Inclusion criteria:

* age 19 years or older
* sustained a TBI
* at least 6-months or greater out from injury
* willing to work on one or more health goals among any of the following areas of focus (e.g., health knowledge, physical activity/exercise, dietary intake/nutrition, stress management, mental activity/stimulation, social ' relationships, leisure, sleep, mindfulness/spirituality, substance use)
* able to potentially participate in physical activity or alter dietary intake, if that is a potential health goal (e.g., no medical contraindication given by their doctor)
* not currently enrolled in a health and wellness program or research study involving a health/wellness program or intervention
* indicates a potential health goal to lose weight and does not independently prepare their own meals, cook, grocery shop, but has a caregiver defined by providing some type of ongoing support (emotional or instrumental) who is willing to participate as a study partner during the intervention condition
* has access to a telephone
* has regular access to the internet from a computer or laptop
* not pregnant (due to the effect on engaging in certain health promoting behaviors such as weight loss)
* does not have a significant psychiatric disorder, such as schizophrenia or bipolar disorder (those with depression or anxiety will not be excluded)

Exclusion criteria:

* non-English speaking
* difficulty hearing
* significant problems with communication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Health Promoting Lifestyle Profile II | Up to 13 months
  HPLP-II; Total scores and subscale scores are summed and divided by number of items on each scale respectively for an average, with higher scores indicating greater lifestyle behaviors

SECONDARY OUTCOMES:
Barriers to Physical Activity and Disability Survey | Up to 13 months
  BPADS: Response choices (yes/no) for 31 items are summarized; 3 items are open-ended, higher scores indicate greater barriers
Social Support and Exercise Support for Eating and Physical Activity Habits | Up to 13 months
  SSES: Subscale scores are obtained for exercise support (ranging from 10 for friends and 10 for family to 80 for friends and 80 for family); higher scores indicate greater support
Stages of Change Readiness and Treatment Engagement Scale | Up to 13 months
  SOCRATES: Items are summed and averaged across each subscale: Recognition scores range from 7-35; Ambivalence scores range from 4-20; Taking Steps scale range from 8-40: Higher scores indicate greater motivation
Patient Health Questionnaire-9 Item | Up to 13 months
  PHQ-9: Scores are summed and range from 0 to 27, higher scores indicate greater depressive symptomatology
Fatigue Severity Scale | Up to 13 months
  FSS: Scores range from 9 to 63 with higher scores indicating greater fatigue
Bodily Pain Index | Up to 13 months
  BPI: Scores for the Interference scale are summed and average for a mean (range 0 to 70) with higher scores indicating greater pain interference
Craig Handicap Assessment Reporting Technique short form | Up to 13 months
  CHARTsf: Suscales scores are summed and averaged for respective scales with higher scores indicating greater community integration
Perceived Wellness Survey | Up to 13 months
  PWS: A total score and subscale scores are calculated with a formula and range between 36 to 316 and average with higher scores indicating greater personal wellness
Barriers to Health Activities among Disabled Persons scale | Up to 13 months
  BHADP: Ratings are summed across each item for how interfering they are with health promotion (range of possible scores 18 to 72)
Zarit Burden Scale | Up to 13 months
  ZBS: Scores are summed (ranges 0 to 48) for a total scores, higher scores are indicative of greater burden
Sociodemographic Characteristics | Up to 13 months
  No abbreviation: Frequencies, summed total, or averages are reported to characterize the sample

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Will need IRB approval